CLINICAL TRIAL: NCT04968704
Title: Computer Modelling Using 2D and 3D Photographs of Patients Faces to Improve Surgical Reconstructive Planning in a Clinical Case Series of Patients With Facial Defects and Improve Patient Satisfaction
Brief Title: Computer Modelling to Plan Surgical Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prateush Singh, NIHR Academic Clinical Fellow, Royal Free Hospital NHS Foundation Trust
Other Study IDs: 299483
Record Dates: First submitted 2021-06-29; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Surgery; Cancer of Skin
Keywords: facial reconstruction; computer modeling; plastic surgery; patient satisfaction
MeSH Terms: conditions — Skin Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — facial skin cancers must be excised- this tissue will be sent to the Royal Free Hospital department of histopathology for review as is standard of care for these patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing facial reconstructive surgery: Patients with facial cancer or disfigurement who require reconstructive surgery will be offered participation in this study.
  Interventions: Other: 3D photography and computer modelling

INTERVENTIONS:
Other: 3D photography and computer modelling — 3D photography is available at our unit department of clinical photography. Photos will be taken and the associated NHS software (Canfield Imaging scientific, inc) used to sit down with the patients and model their reconstruction, thereby reducing anxiety and improving awareness of their treatment plan.

SUMMARY:
The aim of this study is to improve patient satisfaction and outcomes in facial reconstructive surgery by using 3D clinical photography and computer modelling to help illustrate and plan the patients' reconstructive journey.

It will be conducted at the Royal Free Hospital department of Plastic and Reconstructive Surgery, where patients with facial deformities or suspected diagnoses of skin cancer will be referred from their GP or dermatology services. As is routine standard of care, they will be reviewed in outpatient settings and the next management steps initiated. Our study will introduce compulsory 2D and 3D photography and patient satisfaction questionnaires. The photographs will be used to sit down with the participant and illustrate the intended surgical reconstruction, keeping them up to date and fully informed of the surgical plan. The questionnaire, FACE-Q, already validated for facial skin cancer surgery and reconstruction, will be used to assess their satisfaction at each stage of their reconstructive journey.

The results of the study will benefit each participant and illustrate an improvement in satisfaction so that such 3D photography, surgical planning with computer models produced by these 3D images will become a routine part of future patients with facial disfigurement or cancer requiring reconstruction.

This study will form part of a PhD academic qualification at UCL for one of the research registrars.

DETAILED DESCRIPTION:
Setting: Royal Free Hospital, London. Single site. Study Population: Adult patients aged over 18 presenting with;

• Facial defects resulting from cancer or trauma

Consent from the patients will be obtained as soon as possible, during outpatient consultation.

Study design: observational case series, feasibility study. As this is an open observational study, there will be no randomization. As numbers of participant's attending with facial skin cancer defects requiring reconstruction is small, there will not be any sampling.

Expected number of participants: 10. Number determined after discussion with Chief Investigators as adequate to determine feasibility or incorporating 3D photography, computer modelling and questionnaires to improve satisfaction. Statistical input from supervisor and chief investigator, Professor Eva Krumhuber, department of experimental psychology.

Duration of study: 12 months Methodology: Clinic Consultation Patients will be referred to our craniofacial clinic with either pre-defect or pre-biopsy lesions suspicious of being skin malignancies, or following biopsy or defect resulting from excision, trauma or Mohs surgery.

If the lesion is suspicious for cancer but has not been diagnosed, this is discussed with the patient and a biopsy booked. During the consultation the patient is sent for clinical 2D and 3D photography in the Royal Free Hospital Department of Clinical Photography.

If the patient presents to clinic with the defect, multiple pre-defect 2D photographs are requested from the patient and stored on the hospital protected plastic surgery department shared drive.

Photography All patients will undergo outpatient 2D and 3D photography in the Royal Free Hospital Department of Clinical Photography.

Computer modelling All images will be processed using the Vectra XT software from Canfield Imaging Scientific, inc. used at the Royal Free Hospital Department of Clinical Photography. From this, 3D images can be layered, accurate calculations made and the size of defects accurately measured and templated. 3D models can be manipulated to illustrate each stage of the reconstruction.

Treatment modality Treatment modalities will involve standard of care surgical management, pre-assessment and post-operative care. This includes skin cancer and craniofacial MDT multidisciplinary team discussions to plan and decide treatment. This will all take place at Royal Free Hospital, London.

Patient questionnaires Patients will be asked to complete FACE-Q questionnaires at each consultation and after each stage of their reconstruction at initial consultation, 6 weeks post op, 3 months, 6 months and 1 year follow up.

FACE-Q is a validated questionnaire patient reported outcome measure including measures for satisfaction with facial appearance, health-related quality of life, recovery, early life impact, adverse effects and satisfaction with process of care (Klassen et al. 2010).

Follow up For patient who have undergone biopsy, they will be reviewed in the plastic surgery dressings clinic 1 week post op to review the wound; their histology will be discussed in the skin MDT 4-6 weeks later and the patient informed in a consultation of the results.

If further excision or reconstruction is required, the patient will undergo the required imaging and computer modelling and undergo the operative procedure. They will then be reviewed a week later in our dressings clinic and at the next stage of their procedure in 3-4 weeks if staged reconstruction is required. After the final reconstruction, they will be reviewed in outpatient clinic at 6 weeks, 3 months, 6 months and 1 year follow up.

Data collection and storage:

Data will be collected from source (medical notes, questionnaires, and images), and collected on a case record form (CRF) and then transferred to an electronic database. The master database will be recorded by code and will hence be anonymized. Some parts of the medical records and the data collected for the study will be looked at by authorised persons such as the members of the research team, regulatory authorities, the Trust, and the sponsors of this study. They may also be looked at by authorised people to check that the study is being carried out correctly. All will have a duty of confidentiality.

Anonymised extracts of the database may be transferred securely to UCL for analysis. Anonymised images may be shared with researchers in the department of surgery and interventional sciences at UCL.

In some circumstances the data in an anonymous form may be used for preparation of the trial report, and for submission to Government agencies as part of the procedures.

The data may be required for further studies, in which case further Research Ethics Committee approval will be sought. Access to personal data is strictly controlled and limited to authorised personnel only.

Personal data will be stored on paper forms held in a secure, locked office accessible to authorised personnel only. At the end of the study, personal data in paper form (completed Case Record Forms) will be archived securely.

The dataset will be used for the sole purpose set out in this protocol. Anonymised raw data will not be shared with any other organisation or named individual.

In the study, data will be collected from patients in accordance with the patient consent form, patient information sheet and as described in this protocol.

The data will be appropriately maintained by authorised members of the research team for statistical analysis.

The Chief Investigator will nominate an individual to process, store and dispose of study data in accordance with all applicable legal and regulatory requirements, including the Data Protection Act 1998 and any amendments thereto.

Non anonymised data will not be transferred to any party not identified in the protocol and will not be processed and/or transferred other than in accordance with the patients' consent.

ELIGIBILITY:
Inclusion Criteria:

* Participants requiring to undergo facial reconstructive surgery as a result of defects from cancer, trauma or congenital abnormality.
* Participants aged 18 years old or over

Exclusion Criteria:

* If unable to provide written informed consent.
* Younger than 18 years.
* Patients with lesions or defects on the scalp, ears or neck

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with facial skin cancer or disfigurement as a result of trauma or congenital abnormality requiring reconstructive surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
To determine if increasing utilisation of 3D photography and computer modelling in facial reconstructive surgery changes patient satisfaction during their reconstructive journey. | at start of study at at 6 months
  using the validated FACE-Q questionnaire for patients with skin cancer

CONTACTS AND LOCATIONS:
Overall Officials: prateush singh, mbbchir, Principal Investigator — royal free hospital ACF

IPD SHARING:
Plan to Share IPD: No
no data will be shared with researchers outside of the research team